CLINICAL TRIAL: NCT00687206
Title: Efficacy and Safety of Valsartan 160 mg Plus Hydrochlorothiazide 25 mg Once a Day in Patients With Slight Hypertension and Target Organ Damage
Brief Title: Efficacy and Safety of Valsartan Plus Hydrochlorothiazide in Patients With Slight Hypertension and Target Organ Damage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Serafino Fazio MD, Federico II University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Val25/08
Record Dates: First submitted 2008-05-19; First posted 2008-05-30 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Hypertension; Ventricular Remodeling; Erectile Dysfunctions
MeSH Terms: conditions — Hypertension; Ventricular Remodeling; Erectile Dysfunction | interventions — Valsartan; Hematocrit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Valsartan 160mg plus HCT 25mg

INTERVENTIONS:
Drug: Valsartan 160mg plus HCT 25mg — valsartan 160 mg once a day for 6 months plus hydrochlorothiazide 25 mg a tablet once a day for 6 months
  Other Names: Corixil 160/25mg; Cotareg 160/25mg

SUMMARY:
Patients with slight increase in blood pressure levels have an increased cardiovascular risk. In particular this has been demonstrated also in subjects with high-normal blood pressure in whom an exaggerated blood pressure increase, during exercise, and structural left ventricular abnormalities have been shown. On the other hand, the last American and European guidelines for management of hypertension recommend more aggressive treatment in young-middle aged subjects to achieve a better control of cardiovascular risk due to blood pressure increase. In agreement with these recommendations the investigators share the idea that a good blood pressure control should be achieved not only at rest, but also during psycho-physical stress conditions that frequently occur during daily life. On this basis, the investigators decided to evaluate the efficacy and tolerability of the association of valsartan and hydrochlorothiazide (160 an 25 mg daily, respectively) in patients with high-normal blood pressure and first degree arterial hypertension with evidence of organ damage.

The aim of this study is to assess if an early and adequate therapy could bring to a better pressure control (even during physical activity) and a regression of organ damage without interfering with metabolism and erectile function

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65
* Gender Males
* High-normal blood pressure (130-139 mmHg or 85-89 mmHg)
* First degree hypertension (140-159 mmHg or 90-99 mmHg)
* Cardiac remodeling (left ventricular concentric hypertrophy

Exclusion Criteria:

* Coronary artery disease
* Secondary hypertension
* Diabetes mellitus
* Incapacity to perform ergometry test
* Anemia (Hb < 12.5g/dL)
* Cardiac valve disease
* Arrhythmia

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The aim of this study is to assess if an early and adequate therapy could bring to a better pressure control (even during physical activity) and a regression of organ damage assessed by bicycle stress test and mono-bidimensional echocardiography. | 3 and 6 months

SECONDARY OUTCOMES:
Effects of Valsartan 160mg / HCT 25mg on metabolism and erectile function | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Serafino Fazio, MD, Principal Investigator — Federico II University
Locations (1):
- Department of internal medicine University Federico II, Naples, Italy